CLINICAL TRIAL: NCT06936982
Title: Development and Application of a Mechanistic Model and Public Database on Exercise and Health
Brief Title: Research on the Complex Scientific Mechanisms Underlying Exercise and Health: Construction and Application of a Mechanistic Model and Public Database（CISS）
Acronym: CISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aiyoudong Children and Youth Sports Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Basic-2320; 2022YFC3600204 (Other Grant/Funding Number: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus With Dawn Phenomena
MeSH Terms: interventions — Sports Nutritional Physiological Phenomena; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group with a one-day interval (Experimental): A 5-day mini-cycle, with exercise on days 1, 3 and 5, and rest on days 2 and 4. There is an interval of 1 day between mini-weeks.
  Interventions: Other: Sports Exercise
- Group with a two-day interval (Experimental): A 5-day mini-cycle, with exercise on days 1, 3 and 5, and rest on days 2 and 4. There is an interval of 2 day between mini-weeks.
  Interventions: Other: Sports Exercise
- Group with a three-day interval (Experimental): A 5-day mini-cycle, with exercise on days 1, 3 and 5, and rest on days 2 and 4. There is an interval of 3 day between mini-weeks.
  Interventions: Other: Sports Exercise
- Control group (Placebo Comparator): No intervention
  Interventions: Other: control group

INTERVENTIONS:
Other: Sports Exercise — The exercise intervention program used a combination of moderate-intensity aerobic exercise and resistance exercise in the form of exercise day time: 9:00 a.m. to 10:30 a.m., in which 10min warm-up exercise after 45min aerobic exercise, each aerobic exercise 10-12min, with a rest in the middle of the rest 3-5min. resistance exercise was placed in the aerobic exercise after the resistance exercise, resistance exercise using 3 movements, 2 groups, each group 10 times. Each movement was performed 10 times, with a 3-min break between each movement in each group and a 5-min break between groups. 15-min stretching exercises were performed after the exercise. The RPE scale was examined during the exercise, and the subjects were asked about the RPE scale level at the end of every 10 min during the exercise.
  Arms: Group with a one-day interval; Group with a three-day interval; Group with a two-day interval
Other: control group — No intervention
  Arms: Control group

SUMMARY:
Dear Sugar Lovers:

Greetings!

In order to improve the knowledge of chronic disease prevention and control of sugar users and promote health, the investigators plan to organise participants to participate in the Diabetes Exercise Intervention, Science Promotion and Publicity of Chronic Disease Prevention and Control Knowledge Survey, and the investigators hope to get participant's support and cooperation. Please read the following procedure carefully:

1. Exercise intervention: we 2023 late November to start the intervention course.
2. Blood test 2 times (fasting insulin, glycated haemoglobin, total cholesterol, triglyceride, HDL, LDL, fasting blood glucose, tumour necrosis factor, etc., finger blood glucose.

   All the above tests are free of charge
3. popularisation: we will join hands with the community health service centre of Liaojin Village to conduct at least 3 talks on the prevention and control of diabetes.

   The investigators will cooperate with the community health service centre of Lijincun to carry out at least 3 times of knowledge dissemination on diabetes prevention and control.
4. Chronic disease knowledge prevention and control survey: For your physical and mental health development, the follow-up questionnaire is a knowledge survey questionnaire.

Please read the questions carefully. Participants privacy and confidentiality will be strictly protected and will not be disclosed to any unauthorised person.

If participants agree to participate in the programme, please confirm the following information and sign!

1. Co-operation and co-ordination: the investigators promise to participate in the whole project and maintain good communication and co-operation.

   The investigators will keep abreast of and respond to notices, feedback and suggestions, and provide the necessary support and co-operation.
2. Informed Consent: The investigators understand and agree to participate in the project.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM and diagnosed 6 months or more ago
* Meet the criteria of the dawn phenomenon
* Willing to sign the informed consent form
* Voluntarily accept the relevant examinations and tests
* No change in sleep habits in the past 2 weeks

Exclusion Criteria:

* T1DM, special type of diabetes, secondary diabetes, gestational diabetes;
* Nocturnal hypoglycemic reactions due to oral hypoglycemic agents or insulin use
* Patients with serious complications

Ages: 50 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | Approximately 10 weeks from formal enrollment to the end of the intervention
  Blood glucose was tested using a continuous glucose measurement system, which was worn throughout the intervention and allowed the concentration of blood glucose to be tested and recorded every 3 seconds, with a headcount of 93 at the time of limit collection.
  The number of people at the end of the intervention was 85.
Interleukin-6 | Approximately 10 weeks from formal enrollment to the end of the intervention
  Interleukin-6 concentrations at baseline testing, in pg/mL, Number of Participants with 93. Interleukin-6 concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is ng/L.
Interleukin-8 | Approximately 10 weeks from formal enrollment to the end of the intervention
  Interleukin-8 concentrations at baseline testing, in pg/mL, Number of Participants with 93. Interleukin-8 concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is pg/mL.
Tumor necrosis factor-α | Approximately 10 weeks from formal enrollment to the end of the intervention
  Tumor necrosis factor-α concentrations at baseline testing, in pg/mL, Number of Participants with 93. Tumor necrosis factor-α concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is μg/L.
Hypertension | Approximately 10 weeks from formal enrollment to the end of the intervention
  Hypertension concentrations at baseline testing, in pg/mL, Number of Participants with 93. Hypertension concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is mmHg.
Body mass index，BMI | Approximately 10 weeks from formal enrollment to the end of the intervention
Fat content | Approximately 10 weeks from formal enrollment to the end of the intervention
  Measured by Inbody, a body composition tester using bioelectrical impedance, in Kg.
Muscle content | Approximately 10 weeks from formal enrollment to the end of the intervention
  Measured by Inbody, a body composition tester using bioelectrical impedance, in Kg.
Body fat percentage | Approximately 10 weeks from formal enrollment to the end of the intervention
  Measured by Inbody, a body composition tester using bioelectrical impedance, in %.
Superoxide dismutase | Approximately 10 weeks from formal enrollment to the end of the intervention
  Superoxide dismutase concentrations at baseline testing, in pg/mL, Number of Participants with 93. Superoxide dismutase concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is U/mL.
Glutathione peroxidase | Approximately 10 weeks from formal enrollment to the end of the intervention
  Glutathione peroxidase concentrations at baseline testing, in pg/mL, Number of Participants with 93. Glutathione peroxidase concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is U/L.
Total Cholesterol | Approximately 10 weeks from formal enrollment to the end of the intervention
  Total Cholesterol concentrations at baseline testing, in pg/mL, Number of Participants with 93. Total Cholesterol concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is mmol/L.
Triglyceride | Approximately 10 weeks from formal enrollment to the end of the intervention
  Triglyceride concentrations at baseline testing, in pg/mL, Number of Participants with 93. Triglyceride concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is mmol/L.
High-density lipoprotein cholesterol | Approximately 10 weeks from formal enrollment to the end of the intervention
  High-density lipoprotein cholesterol concentrations at baseline testing, in pg/mL, Number of Participants with 93. High-density lipoprotein cholesterol concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is mmol/L.
Low-Density Lipoprotein Cholesterol | Approximately 10 weeks from formal enrollment to the end of the intervention
  Low-Density Lipoprotein Cholesterol concentrations at baseline testing, in pg/mL, Number of Participants with 93. Low-Density Lipoprotein Cholesterol concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is mmol/L.
Glycosylated Hemoglobin, Type A1c | Approximately 10 weeks from formal enrollment to the end of the intervention
  Glycosylated Hemoglobin, Type A1c concentrations at baseline testing, in pg/mL, Number of Participants with 93. Glycosylated Hemoglobin, Type A1c concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is mmol/L.
△Damw | Approximately 10 weeks from formal enrollment to the end of the intervention
  △Damw(mmol/L)=FBG-Lowest blood sugar at night
Fasting insulin | From enrollment to the end of intervention at 10 weeks
  Fasting insulin concentrations at baseline testing, in pg/mL, Number of Participants with 93. Fasting insulin concentration 24 hours after the end of the intervention, Number of Participants with 85. The unit is μIU/mL.
HOMA-β | Approximately 10 weeks from formal enrollment to the end of the intervention
  HOMA-β=20×［FINS(IU/mL)］/［FBG(mmol/L)-3.5］(%)
HOMA-IR | Approximately 10 weeks from formal enrollment to the end of the intervention
  HOMA-IR=［FBG(mmol/L)×［FINS (mIU/L)］/22.5
ISI | Approximately 10 weeks from formal enrollment to the end of the intervention
  ISI=1/［FBG(mmol/L)×FINS (mIU/L)］

CONTACTS AND LOCATIONS:
Locations (1):
- Suojincun Community Health Service Center, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of the subjects.